CLINICAL TRIAL: NCT07164326
Title: Dexmedetomidine Nebulization for Attenuation of Pressor Response to Laryngoscopy and Endotracheal Intubation in Sever Preeclamptic Patients Undergoing Caesarean Section Under General Anaesthesia
Brief Title: Dexmedetomidine Nebulization for Attenuation of Pressor Response to Laryngoscopy and Endotracheal Intubation in Sever Preeclamptic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Sayed Hussein Hassan, Dexmedetomidine nebulization for attenuation of pressor response to laryngoscopy and endotracheal intubation in sever preeclamptic patients undergoing caesarean section under general anaesthesia. A prospective randomized clinical trial., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dexmedetomidine nebulization
Record Dates: First submitted 2025-08-30; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Pressor Response
Keywords: Preeclampsia; Nebulization
MeSH Terms: conditions — Pre-Eclampsia | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental): Nebulization of dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- Saline (Placebo Comparator): Nebulization of saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Nebulization of dexmedetomidine
  Arms: Dexmedetomidine
Drug: Saline — Nebulization of normal saline
  Arms: Saline

SUMMARY:
Dexmedetomidine nebulization in sever preeclamptic patients

DETAILED DESCRIPTION:
Dexmedetomidine nebulization for attenuation of pressor response to laryngoscopy and endotracheal intubation in sever preeclamptic patients undergoing caesarean section under general anaesthesia. A prospective randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe pre-eclampsia scheduled for cesarean section under general anesthesia
* ASA II, III

Exclusion Criteria:

* sever obesity (BMI ≥ 40)
* Cardiac patients
* History of diabetes mellitus
* Renal dysfunction (elevated serum creatinine > 2mg\dl)
* hepatic dysfunction (elevated hepatic enzyme three times above normal)
* History to hypersensitivity to the tested drug.
* Emergency surgery
* Known fetal anomalies

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure in response to endotracheal intubation | Intraoperative
  the change in systolic blood pressure in response to endotracheal intubation

SECONDARY OUTCOMES:
Optic nerve sheath diameter | Intraoperative
  the change in optic nerve sheath diameter in response to endotracheal intubation
Incidence of maternal postoperative sore throat | 1 hour Postoperative
Incidence of maternal postoperative hoarseness of voice | 1 hour Postoperative